CLINICAL TRIAL: NCT00605488
Title: Pilot Study Investigating the Biodistribution and Potential Diagnostic Ability of 18F FACBC in Patients With Head and Neck, Breast, and Prostate Cancer
Brief Title: The Biodistribution and Potential Diagnostic Ability of 18F FACBC in Patients With Head and Neck, Breast, and Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-040
Record Dates: First submitted 2008-01-17; First posted 2008-01-31 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Head and Neck Cancer; Prostate Cancer
Keywords: Pet Scan
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Prostatic Neoplasms

ARMS (1):
- 1 (Experimental): Pet Scan
  Interventions: Procedure: novel PET tracer FACBC

INTERVENTIONS:
Procedure: novel PET tracer FACBC — Two IV catheters (heplock) will be placed in your forearms for injection of the dye-like material (FACBC) and blood sampling. An IV blood sample and a urine sample will be taken for testing. These samples will be used to measure the dye, FACBC, in blood and urine. You will be placed in the PET machine, where FACBC will be injected slowly over 30 seconds. Pictures of one region of your body will be taken for up to 60 minutes. Depending on your condition, your actual picture time may be shorter. You will come out of the scanner to stretch, walk around or sit in a chair. An optional urine sample and an IV blood sample will also be taken at this time. Again, these samples will be used to measure the dye, FACBC, in blood and urine. This will be followed by a picture of your body from the neck to the upper thighs. This picture will take about 30 minutes.

SUMMARY:
See where the dye-like material (FACBC) goes in your body and how long it stays in your body. See how much of the dye-like material is picked up by your tumor Compare the FACBC pictures with other pictures (such as FDG PET scan) that were obtained as part of your standard imaging evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ or equal 18 years old
* Scheduled for treatment at Memorial Hospital
* Primary HNSCC or primary breast cancer; histological confirmation of diagnosis at Memorial hospital
* Large primary HNSCC cancer (loco-regional advanced, ≥ or equal to T2) by CT/MRI imaging or clinical exam, without prior treatment, N1-N3
* Large primary breast cancer (≥ or equal to T2) by imaging or clinical impression based physical exam; patients with suspicion of axillary nodal disease (N1-2), without prior treatment
* Established progressive metastatic prostate cancer
* This diagnosis may be based upon histologic confirmation of metastatic disease by biopsy of a lesion OR clear clinical evidence for metastatic disease (e.g., based on clinical findings, laboratory data and/or imaging findings in CT, MRI, or bone scan), as defined by the referring oncologist
* Progressive disease is defined as clear progression on imaging studies (increase in size and number of lesions on bone scan, CT, or MRI) and consecutive rises in PSA as used in clinical management by the prostate cancer oncology group at MSKCC
* FDG PET scan was obtained as part of the clinical work-up, within 4 weeks prior to enrollment. This clinical FDG PET scan should be done at MSKCC.
* Disease can be clearly demonstrated by structural imaging (CT or MRI) or bone scan. This may include characteristic bone lesions on bone scan, CT or MRI; AND/OR measurable soft tissue/nodal lesions on CT or MRI.
* Minimum tumor/metastasis size of 1 cm
* Negative pregnancy test

Exclusion Criteria:

* Patient cannot tolerate lying still for approximately 60 minute sessions in the PET tomograph.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-04-25; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
To study the biodistribution and dosimetry of FACBC in patients with head and neck squamous cell carcinoma (HNSCC), breast cancer and prostate cancer. | conclusion of study

SECONDARY OUTCOMES:
To compare these FACBC data with PET imaging findings using the current clinical standard PET tracer FDG. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org